CLINICAL TRIAL: NCT01719536
Title: Conmana Versus Pemetrexed-based First-line Induction and Maintenance Chemotherapy in Advanced Lung Adenocarcinoma With EGFR-mutation
Brief Title: Icotinib Versus First-line Chemotherapy Plus Maintenance Treatment in EGFR Positive Lung Adenocarcinoma Patients
Acronym: Convince
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV36
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: NSCLC
MeSH Terms: interventions — icotinib; Drug Therapy; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Icotinib (Experimental): Icotinib 125mg is administered orally three times per day.
  Interventions: Drug: Icotinib
- Chemotherapy (Active Comparator): Patients in this arm will receive pemetrexed/cisplatin for 4 cycles, of who don't progress will receive maintenance treatment with pemetrexed.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Icotinib — Icotinib: 125 mg is administered orally three times per day.
  Other Names: BPI-2009; Conmana
  Arms: Icotinib
Drug: Chemotherapy — First-line chemotherapy: pemetrexed/cisplatin for 4 cycles. Maintenance treatment: pemetrexed.
  Other Names: ALIMTA
  Arms: Chemotherapy

SUMMARY:
The purpose of this study is to compare icotinib with induction and maintenance chemotherapy in the first-line treatment of advanced non-small cell lung cancer (NSCLC) patients with EGFR mutation.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of icotinib and pemetrexed-based first-line induction and maintenance chemotherapy in advanced lung adenocarcinoma with EGFR-mutation，primary endpoint is progress-free survival，second endpoints include overall survival, time to progression, and so on.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or progressive Non-Small Cell Lung Cancer stage IV or IIIB patients.
* Positive EGFR Mutation.
* No previous systemic anticancer therapy.
* Measurable lesion according to RECIST with at least one measurable lesion not previously irradiated, unless disease progression has been documented at that site.
* Provision of written informed consent.

Exclusion Criteria:

* Experience of Anti-EGFR(the epidermal growth factor receptor) Monoclonal Antibody or small molecular compounds therapy such as gefitinib, erlotinib or Cetuximab.
* Evidence of clinically active Interstitial Lung Diseases (Patients with chronic, stable, radiographic changes who are asymptomatic need not be excluded).
* Known severe hypersensitivity to icotinib or any of the excipients of this product.
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2012-12; Primary Completion 2016-09 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 12 months
  A duration from randomization date to disease progression(as defined by RECIST) or death. If a participant are known to have progressed, the time to progression is defined as the time from the date of randomization to the date of progression. Otherwise, a participant will be censored at the last date they are known not to be progressed.

SECONDARY OUTCOMES:
Overall survival | 20 months
  Overall Survival is assessed via calculation of the time to death due to any cause. If a participant is known to have died, the time to death is defined as the time from the date of randomization to the date of death. Otherwise, a participant will be censored at the last date they are known to be alive.
Objective response rate | 12 weeks
  Number of participants who achieve complete response or partial response. Either complete response (CR) or partial response (PR) will be evaluated by RECIST, confirmed at least 28 days following the date of the initial response.

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuankai, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (21):
- China (21):
  - The First Affiliated Hospital of Anhui Medical Univercity, Hefei, Anhui
  - Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality
  - Beijing Hospital for Chest Tumors & Tuberculosis Diseases, Beijing, Beijing Municipality
  - Xinqiao Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Guangzhou Medical Collage, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Hebei Provincal Tumor Hospital, Shijiazhuang, Hebei
  - Harbin Medical Univercity Cancer Hospital, Harbin, Heilongjiang
  - Henan Provincal Tumor Hospital, Zhengzhou, Henan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Provincal Tumor Hospital, Nanjing, Jiangsu
  - The First Bethune Hospital of Jilin Univercity, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Chest Hospital Affiliated to Shanghai Jiaotong Univercity, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan Univercity, Shanghai, Shanghai Municipality
  - Changhai Hospital, The Second Military Medical University, Shanghai, Shanghai Municipality
  - Xijing Hospital, Xian, Shanxi
  - Sichuan Provincal Tumor Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Result] Shi YK, Wang L, Han BH, Li W, Yu P, Liu YP, Ding CM, Song X, Ma ZY, Ren XL, Feng JF, Zhang HL, Chen GY, Han XH, Wu N, Yao C, Song Y, Zhang SC, Song W, Liu XQ, Zhao SJ, Lin YC, Ye XQ, Li K, Shu YQ, Ding LM, Tan FL, Sun Y. First-line icotinib versus cisplatin/pemetrexed plus pemetrexed maintenance therapy for patients with advanced EGFR mutation-positive lung adenocarcinoma (CONVINCE): a phase 3, open-label, randomized study. Ann Oncol. 2017 Oct 1;28(10):2443-2450. doi: 10.1093/annonc/mdx359. PMID 28945850